CLINICAL TRIAL: NCT06902428
Title: A Multi-center, Randomised, Double-blind, Placebo-controlled Phase II Clinical Study Evaluating the Efficacy and Safety of HSK44459 Tablets in Patients With Behçet's Disease
Brief Title: Evaluating the Efficacy and Safety of of HSK44459 in Patients With Behçet's Disease
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSK44459-202
Record Dates: First submitted 2025-03-17; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Behcet's Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): In treatment period, subject will take placebo matching HSK44459 twice daily in the morning and in the evening for 12 weeks. The administration time of the drug should be relatively fixed every day.
  Interventions: Drug: Placebo
- HSK44459 dose 1 (Experimental): In treatment period, subject will take higher dose of HSK44459 twice daily in the morning and in the evening for 12 weeks. The administration time of the drug should be relatively fixed every day.
  Interventions: Drug: HSK44459
- HSK44459 dose 2 (Experimental): In treatment period, subject will take lower dose of HSK44459 twice daily in the morning and in the evening for 12 weeks. The administration time of the drug should be relatively fixed every day.
  Interventions: Drug: HSK44459

INTERVENTIONS:
Drug: HSK44459 — HSK44459, bid p.o.
  Arms: HSK44459 dose 1; HSK44459 dose 2
Drug: Placebo — Placebo, bid p.o.
  Arms: Placebo

SUMMARY:
This is a phase 2, multi-center, randomised, double-blind, placebo-controlled study with an equal randomization among the HSK44459 dose 1, dose 2 and placebo treatment groups. The main objective is to evaluate of the efficacy and the secondary objective is to evaluate the safety and pharmacokinetic.

DETAILED DESCRIPTION:
This study is a phase 2, multi-center, randomized, double - blind, placebo - controlled study designed to evaluate the efficacy and safety of HSK44459 in the treatment of patients with Behçet Disease (BD). Approximately 120 subjects will be randomized into this study.

The entire study will consist of 3 phases: a screening phase, a 12-week treatment phase, and a 4-week follow-up phase.

Screening: All subjects will undergo a screening period of up to 6 weeks before the first dose (Visit 3, Day 1).

Treatment phase: Eligible BD patients will be randomly assigned to the HSK44459 dose 1 group, the HSK44459 dose 2 group, or the placebo group. During the treatment period, HSK44459 or placebo will be administered twice daily for 12 weeks.

Follow-up phase: Subjects in the study (including those who withdraw from treatment for any reason) will have an additional 4 - week follow-up after the end of the last administration.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged between 18 and 75 years (inclusive) at the time of signing the informed consent document.
2. Diagnosed with Behçet's disease (BD) meeting the International Criteria for Behçet's Disease (ICBD, ICBD-2013) criteria.
3. Suffered from at least 3 episodes of oral ulcers within 12 months prior to randomization.
4. Had at least 2 oral ulcers present during the Screening Phase.
5. Had received drug treatment for Behçet's disease.
6. Eligible for systemic treatment of oral ulcers.
7. Consented to participate in this trial, and voluntarily signed the informed consent form.

Exclusion Criteria:

1. Active involvement of major organs related to Behçet's disease - pulmonary (eg, pulmonary artery aneurysms), vascular (eg, thrombophlebitis), gastrointestinal (eg, gastrointestinal ulcers), and central nervous system (eg, meningoencephalitis) manifestations, and ocular lesions (eg, uveitis) requiring immunosuppressive treatment.
2. Subjects who have received the following immunomodulatory treatments, including:

   1. Hydroxychloroquine was used within 5 days prior to randomization;
   2. Colchicine was used within 7 days prior to randomization;
   3. Azathioprine, mycophenolate mofetil, baricitinib, or tofacitinib was used within 10 days prior to randomization;
   4. Cyclosporine, methotrexate, cyclophosphamide, thalidomide, or dapsone was used within 4 weeks (28 days) prior to randomization;
   5. Biological agents were used within 5 half-lives prior to randomization;
3. Subjects who have received systemic corticosteroid treatment prior to randomization;
4. Subjects who have used traditional Chinese patent medicines with immunomodulatory effects within 2 weeks prior to randomization; those who have taken traditional Chinese patent medicines that may affect the efficacy within 2 weeks prior to randomization;
5. Patients who have previously received systemic treatment with phosphodiesterase 4 (PDE4) inhibitors;
6. Patients who have used a strong CYP3A4 inhibitor or inducer within 14 days prior to randomization or within 5 pharmacokinetic half-lives (whichever is longer); and patients who insist on taking a strong CYP3A4 inhibitor or inducer during the study period;
7. Subjects who have used any investigational medicinal product within 4 weeks prior to randomization or within 5 pharmacokinetic half-lives (whichever is longer);
8. Laboratory tests during the screening period:

   * Hemoglobin ≤ 90g/L;
   * White blood cell count < 3.0×10⁹/L or white blood cell count > 14×10⁹/L;
   * Platelets < 100×10⁹/L;
   * Estimated Glomerular Filtration Rate (eGFR) ≤ 45 ml/min/1.73 m²;
   * Total bilirubin > 1.5×ULN;
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) are both > 1.5×ULN;
9. Subjects with clinically significant abnormalities in chest X-ray or CT examination at the time of screening, and as judged by the investigator, may place the subject at safety risk;
10. Subjects with a history of active or recurrent bacterial, viral, fungal, mycobacterial, or other infections (including but not limited to tuberculosis and atypical mycobacteriosis, hepatitis B and C, and herpes zoster, but excluding onychomycosis) at the time of screening, or any episode of severe infection within 4 weeks prior to screening that required hospitalization or treatment with intravenous or oral antibiotics;
11. Subjects with other autoimmune diseases or immune-related chronic inflammatory diseases at the time of screening, such as rheumatic fever, rheumatoid arthritis, systemic lupus erythematosus, etc.;
12. Subjects who have undergone or plan to undergo major surgery (evaluated as major surgery by the investigator) within 3 months prior to screening or during the study period;
13. Subjects whose blood pressure was still not controlled after treatment with antihypertensive drugs within 3 months prior to screening, and whose blood pressure was ≥ 160/100 mmHg during the screening period;
14. Subjects who had a thromboembolic event (including stroke and transient ischemic attack) within 6 months prior to screening;
15. Subjects who had any clinically significant heart disease (such as but not limited to unstable ischemic heart disease, NYHA class III/IV left ventricular failure, or myocardial infarction) discovered within 6 months prior to screening or those with clinically significant 12-lead electrocardiogram abnormalities, and as judged by the investigator, may place the subject at safety risk or may interfere with the study evaluation;
16. Subjects with a history of attempted suicide within 2 years prior to screening, or a history of major psychiatric illness requiring hospitalization within 3 years prior to screening;
17. Subjects with a history of malignant tumor within 5 years prior to screening (except for patients with treated basal cell carcinoma of the skin, in situ squamous cell carcinoma of the skin, or in situ cervical cancer);
18. History of gastrointestinal surgery or diseases (excluding appendectomy or simple hernia repair) that may interfere with the pharmacokinetics (PK) of the investigational drug;
19. Subjects with active hepatitis B (positive for hepatitis B surface antigen (HBsAg) and hepatitis B virus DNA (HBV-DNA) higher than the upper limit of the normal range), positive for hepatitis C antibody, syphilis infection (positive for anti-TP test), or human immunodeficiency virus (HIV) infection (positive for anti-HIV) during the screening period;
20. Subjects with a history of drug abuse, drug use, or excessive alcohol consumption within 3 months prior to screening. Excessive alcohol consumption means an average daily alcohol intake of > 2 units of alcohol;
21. Subjects with a history of severe drug allergy or those allergic to the investigational medicinal product specified in the protocol;
22. Pregnant and lactating women, or women who plan to become pregnant or breastfeed during the study period;
23. Subjects whom the investigator deems to have any other factors that make them unsuitable for participating in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03-24 (Estimated); Primary Completion 2026-06-05 (Estimated); Study Completion 2026-07-03 (Estimated)

PRIMARY OUTCOMES:
Area Under the Curve for the Number of Oral Ulcers From Baseline Through treatment period. | 12 weeks
  For the analysis of the primary endpoint, the count of oral ulcers included both existing and recurrent ulcers at each time point.

SECONDARY OUTCOMES:
Percentage of Participants Who Experienced an Oral Ulcer Complete Response at Week 12 | 12 weeks
  A complete response at week 12 was defined as participants being free of oral ulcers at that time point.
Baseline in Oral Ulcer Pain as Measured by Visual Analog Scale at Week 12 | 12 weeks
  The pain of oral ulcers was gauged via a 100-millimeter Visual Analog Scale. Participants were instructed to mark a single perpendicular line across the VAS at a position that corresponded to the intensity of their oral-ulcer pain experienced in the preceding 2 weeks. On this scale, 0 mm (the left-hand extremity) signified the absence of pain, while 100 mm (the right-hand extremity) represented the most excruciating pain one could envision. The measurement from the left-hand end of the scale to the perpendicular line was documented.
Percentage of Participants Who Experienced a Complete Response For Genital Ulcers at Week 12 | 12 weeks
  A complete response at week 12 was defined as participants being free of genital ulcers at that time point.
Change From Baseline in Genital Ulcer Pain as Measured by VAS Score at Week 12 | 12 weeks
  The pain of genital ulcers was gauged via a 100-millimeter Visual Analog Scale. Participants were instructed to mark a single perpendicular line across the VAS at a position that corresponded to the intensity of their genital-ulcer pain experienced in the preceding 2 weeks. On this scale, 0 mm (the left-hand extremity) signified the absence of pain, while 100 mm (the right-hand extremity) represented the most excruciating pain one could envision. The measurement from the left-hand end of the scale to the perpendicular line was documented.
Change From Baseline in Disease Activity as Measured by Behçet's Disease Current Activity Form (BDCAF) at Week 12 | 12 weeks
  The Behçet's Disease Current Activity Form (BDCAF) is composed of three component scores, namely the Behçet's Disease Current Activity Index (BDCAI) score, the Patient's Perception of Disease Activity, and the Clinician's Overall Perception of Disease Activity. The BDCAI encompasses 12 questions that focus on disease manifestations occurring within the past 4 weeks. These manifestations include the activity of oral and genital diseases, along with other symptoms of Behçet's Disease (BD) affecting the skin, joints, gastrointestinal (GI) tract, eyes, nervous system, and vascular system. The BDCAI score is calculated as the sum of the scores for these 12 items and can range from 0 to 12. A higher score on the BDCAI indicates a more severe level of disease activity (i.e., the condition is worsening).
Change From Baseline in Disease Activity as Measured by Behçet's Syndrome Activity Score (BSAS) at Week 12 | 12 weeks
  The Behçet's Syndrome Activity Score (BSAS) is composed of 10 questions that assess the number of new oral and genital ulcers and skin lesions, GI, CNS, vascular, and ocular involvement, and the participant's current level of discomfort. The Behçet's Syndrome Activity Score spans from 0 to 100. A higher score on this scale corresponds to a more severe level of disease activity. When there is a decrease in the score compared to the baseline value, it indicates an improvement in the patient's condition.
Change From Baseline in Behçet's Disease Quality of Life (BD Qol) Scores at Week 12 | 12 weeks
  The Behçet's Disease Quality of Life (BDQoL) questionnaire was designed to assess the impact of Behçet's disease on a participant's daily life. It includes 30 self-administered questions that evaluate the limitations imposed by the disease on the participant's activities and their emotional reactions to these limitations. The overall score is calculated by summing the responses to all 30 items, where each "yes" response is scored as 1 and each "no" response as 0. A total score of 0 indicates no effect of Behçet's disease on the participant's quality of life, while a score of 30 reflects the most significant impact. A decrease in the score from baseline signifies an improvement in the participant's quality of life.
Change From Baseline in Quality of Life as Measured by Short Form 36 Health Survey | 12 weeks
  The SF-36 is a validated, self-administered 36-item general health status instrument often used in clinical trials and health services research. It consists of 8 scales: physical function (PF), role-physical (RP), vitality (VT), general health (GH), bodily pain (BP), social function (SF), role-emotional (RE), and mental health (MH).
Time to Oral Ulcer Complete Response | 12 weeks
  The time to complete response of oral ulcers was defined as the interval from the date of the first dose to the date when a complete response was first attained during the treatment phase.
Percentage of Participants Exhibiting No Oral Ulcers After a Complete Response | 12 weeks
  The definition encompasses participants who, subsequent to achieving a complete response (characterized by the absence of oral ulcers) prior to week 12, maintained an oral ulcer-free status throughout the entirety of the period up to and including week 12.
Percentage of Participants Who Achieved an Oral Ulcer Complete Response at Week 6 and Remained Oral Ulcer-Free for at Least 6 Additional Weeks | 12 weeks
  Participants who were oral ulcer-free at week 6 and maintained an oral ulcer-free status throughout the entirety of the period up to and including week 12.
Number of recurrences of oral ulcers after complete response through week 12 | 12 weeks
  The number of oral ulcers reported upon the initial loss of complete response. This refers to the first occurrence where, subsequent to achieving complete response, a participant experiences a recurrence of oral ulcers during the treatment phase.
The incidence rate and severity of adverse events | 16 weeks
  An Adverse Event (AE) refers to all adverse medical events that occur to subjects in a clinical study. It can manifest as symptoms/signs, diseases, or abnormal laboratory test results, but it is not necessarily causally related to the investigational medicinal product. In this study, all adverse events that occur from the time of signing the informed consent form until the end of the safety follow-up period will be recorded.
Maximum Plasma Concentration (Cmax) | 12 weeks
  the population pharmacokinetic (popPK) characteristics Cmax of HSK44459 in subjects
Elimination half-life (T1/2) | 12 weeks
  the population pharmacokinetic (popPK) characteristics T1/2 of HSK44459 in subjects
Area under drug time curve (AUC) | 12 weeks
  the population pharmacokinetic (popPK) characteristics AUC of HSK44459 in subjects